CLINICAL TRIAL: NCT00140855
Title: A Phase II Study of Anti-CTLA-4 Antibody in Advanced Synovial Sarcoma Patients
Brief Title: A Study of Anti-CTLA-4 Antibody in Patients With Advanced Synovial Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study discontinued due to poor accrual.
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Medarex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2002-010; MSKCC 04-128 (Other: MSKCC)
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2021-07-14 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Synovial Sarcoma
Keywords: synovial sarcoma; immunotherapy; cancer-testis antigen; cancer-germ cell antigen; soft tissue sarcoma; SYT-SSX chromosomal translocation
MeSH Terms: conditions — Sarcoma, Synovial; Sarcoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ipilimumab (Experimental): Three doses of ipilimumab, 3 mg/kg, were administered by intravenous infusion at 3-week intervals. A 6-week observation period followed the final dose.
  Interventions: Biological: ipilimumab

INTERVENTIONS:
Biological: ipilimumab
  Other Names: Anti-CTLA-4 monoclonal antibody; monoclonal antibody MDX-010; Yervoy

SUMMARY:
The purpose of this study is to determine whether immune therapy with anti-CTLA-4 antibody is effective in people with advanced synovial sarcoma.

DETAILED DESCRIPTION:
Approximately 750-900 people in the United States each year develop synovial sarcoma, a rare form of cancer of connective tissue. This tumor frequently metastasizes to other parts of the body such as the lungs. Chemotherapy can sometimes decrease the size of the recurrent tumors, but these results are usually only temporary, and the tumors grow again.

We are trying to exploit some of the proteins made by synovial sarcoma (cancer-germ cell or cancer-testis antigens) as targets for the immune system. Specifically, we are investigating if immune-based therapy with anti-CTLA-4 antibody once every 3 weeks for three treatments will activate the immune system enough to attack recurrent synovial sarcoma. In this study the tumor itself serves as the "vaccine" or source of protein, as we try to activate tumor-fighting T cells with the anti-CTLA-4.

Anti-CTLA-4 takes the brakes off the immune system to allow otherwise hidden immune responses to become more active. In so doing, there could be other side effects, such as immune system attacks against the normal organs of the body. We will follow both the anti-tumor immune responses with frequent blood tests and follow and treat side effects people develop on this study to determine if anti-CTLA-4 is worth pursuing in a larger number of patients with synovial sarcoma or other sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented synovial sarcoma.
* Patients with metastatic disease or locally recurrent disease who have failed or refused standard treatment. The disease must be measurable by RECIST.
* Expected survival of at least 6 months.
* Weight at least 35 kg.
* ECOG performance scale 0-2.
* At least 3 weeks since major surgery, and at least 3 weeks since completing radiation therapy or chemotherapy (6 weeks for patients receiving mitomycin C).
* Resolution of toxicity from previous treatment to NCI-CTC grade 1 or less before treatment.
* Adequate bone marrow, renal and hepatic function.
* Able and willing to give valid written informed consent.

Exclusion Criteria:

* Clinically significant heart disease (NYHA Class III or IV).
* Other serious illnesses, e.g. serious infections requiring antibiotics or bleeding disorders.
* History of autoimmune disease.
* Serious intercurrent illness, requiring hospitalization.
* Patients with a second cancer diagnosis in the last five years, except for basal cell carcinoma, completely resected, or cervical carcinoma in situ (CIN), completely resected.
* Known HIV positivity.
* Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may be available.
* Chronic use of immunosuppressive drugs such as systemic corticosteroids.
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
* Lack of availability for immunological and clinical follow-up assessments.
* Participation in any other clinical trial involving another investigational agent within 3 weeks prior to enrollment.
* Pregnancy or breast feeding.
* Refusal or inability to use effective means of contraception (all men, and women with childbearing potential).

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-06-08 (Actual); Primary Completion 2007-04-18 (Actual); Study Completion 2007-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Maki, MD PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Result] Maki RG, Jungbluth AA, Gnjatic S, Schwartz GK, D'Adamo DR, Keohan ML, Wagner MJ, Scheu K, Chiu R, Ritter E, Kachel J, Lowy I, Old LJ, Ritter G. A Pilot Study of Anti-CTLA4 Antibody Ipilimumab in Patients with Synovial Sarcoma. Sarcoma. 2013;2013:168145. doi: 10.1155/2013/168145. Epub 2013 Feb 27. PMID 23554566
- See also: Link to MSKCC Sarcoma Clinical trial web site highlighting anti-CTLA4 protocol — http://www.mskcc.org/mskcc/html/2270.cfm?peds=no&team=Soft+Tissue+Sarcoma&x=18&y=19

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ipilimumab
Started | 6
Completed | 4
Not Completed | 2
Not completed — Progressive disease | 2

BASELINE CHARACTERISTICS:
Population: All subjects who entered the study.
Arm/Group | Ipilimumab
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Best Tumor Response as Measured by the Response Evaluation Criteria in Solid Tumors (RECIST).
Description: Computed tomography (CT) scans were performed at screening, and week 10. Response was assessed using RECIST version 1.0 (Therasse P et al. J Natl Cancer Inst 92:205-216). Per RECIST, target lesions are categorized as follows: complete response (CR): disappearance of all target lesions (no evaluable disease); partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria.
Time Frame: up to 10 weeks
Population: All subjects who entered the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 6
Participants
  CR | 0
  PR | 0
  SD | 0
  PD | 6

2. Secondary Outcome: Number of Subjects With NY-ESO-1 Specific Immunity as Measured by Antibody Response to NY-ESO-1 or LAGE-1
Description: Blood samples were taken at baseline and weeks 4, 7, 10 and 13. Humoral immunity was assessed by measurement of antibodies to NY-ESO-1 or LAGE by enzyme-linked immunosorbent assay (ELISA). Positive results are reported as antibodies to NY-ESO-1- and/or LAGE-1-specific Total IgG (reciprocal titer).
Time Frame: up to 13 weeks
Population: All subjects who entered the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 6
Participants
  Number of subjects with positive antibody titers | 0
  Number of patients with negative antibody titers | 6

3. Secondary Outcome: Number of Subjects Reporting Adverse Events (AEs)
Description: All adverse events (AEs) which occurred after signed informed consent were documented in the source records and on the respective AE Case Report Form (CRF). Toxicity was graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Scale (Version 3.0).
Time Frame: up to 13 weeks
Population: All subjects who entered the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: up to 13 weeks
Description: All adverse events (AEs) which occurred after signed informed consent were documented in the source records and on the respective AE Case Report Form (CRF). Toxicity was graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Scale (Version 3.0).
Groups:
- Ipilimumab: Three doses of ipilimumab 3 mg/kg, were administered by intravenous infusion at 3 week intervals. A 6-week observation period followed the final dose.
Arm/Group | Ipilimumab
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=6)
Lymphopenia (Blood and lymphatic system disorders) | 2
Hyperglycemia (Endocrine disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 3
Bronchitis (Infections and infestations) | 1
Blood alkaline phosphatase (Investigations) | 3
Alanine aminotransferase (Investigations) | 1
Platelet count (Investigations) | 2
Hemoglobin (Investigations) | 1
White blood count (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Chest pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneform (Skin and subcutaneous tissue disorders) | 1
Blood creatinine (Investigations) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Aspartate aminotransferase (Investigations) | 1

LIMITATIONS AND CAVEATS:
This study was terminated early due to slow recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No